CLINICAL TRIAL: NCT02395809
Title: Randomized Clinical Trial of Transcutaneous Electrical Posterior Tibial Nerve Stimulation Versus Lateral Internal Sphincterotomy for Treatment of Chronic Anal Fissure.
Brief Title: Transcutaneous Posterior Tibial Nerve Stimulation for Treatment of Chronic Anal Fissure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Tamer Youssef Mohamed, Tamer Youssef, Mansoura University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MFM201215
Record Dates: First submitted 2015-03-09; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Anal Fissure
MeSH Terms: interventions — Lateral Internal Sphincterotomy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LIS group (Active Comparator): Lateral internal shincterotomy: A blade knife (No 11) was inserted between internal and external sphincter. The tip of the blade was angled medially pointing just above the dentate line and IS was divided. When the knife was felt beneath the intact mucosa, it was withdrawn.
  Interventions: Procedure: lateral internal sphincterotomy
- TENS group (Active Comparator): Posterior tibial nerve stimulation by transcutaneous electrical nerve stimulation by through a stimulating TENS unit.
  Interventions: Procedure: TENS

INTERVENTIONS:
Procedure: lateral internal sphincterotomy
  Arms: LIS group
Procedure: TENS
  Arms: TENS group

SUMMARY:
Lateral internal sphinterotomy (LIS) is the gold standard against which all treatments are compared with a healing rate over 92%. However, the most serious complication of this procedure is anal incontinence. To overcome these problems, continued efforts are being tried to find less invasive treatments modalities for anal fissure that is as effective as surgical therapy with lower morbidity.

DETAILED DESCRIPTION:
Sacral nerve stimulation has been recently tried for management of chronic anal fissure with promising results. However, the technique described is invasive with the need for surgically implantable expensive stimulator electrodes.

The aim of this study was to evaluate the efficacy of posterior tibial nerve stimulation (PTN) by transcutaneous electrical nerve stimulation (TENS) and to compare it to the conventional LIS. This non-invasive technique has been proved to be of acceptable results in treatment of fecal incontinence and urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive symptomatic adults affected by chronic anal fissure were enrolled in the study.

Exclusion Criteria:

1. patients younger than 18 years;
2. patients with laterally located or painless fissures;
3. concurrent fistula or significant hemorrhoidal disease;
4. inflammatory bowel disease;
5. Diabetes mellitus;
6. pregnancy;
7. neurological disease;
8. spinal cord lesions,
9. use of cardiac pacemaker. Males and females were considered for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
number of patients with clinical improvement of symptoms | one year
  Resolution of anal pain after the procedure

SECONDARY OUTCOMES:
number of patients with post-procedure anal incontinence according to Pescatory grading and scoring index for anal incontinence | one year
Number of patients with improvement of constipation according to Wexner constipation score | one year
Anal pain scores on VAS | one month
Post-procedure patient satisfaction on VAS | one year
Number of patients with healed anal fissure | one month
  Complete epithelialization of the fissure

REFERENCES:
- [Derived] Youssef T, Youssef M, Thabet W, Lotfy A, Shaat R, Abd-Elrazek E, Farid M. Randomized clinical trial of transcutaneous electrical posterior tibial nerve stimulation versus lateral internal sphincterotomy for treatment of chronic anal fissure. Int J Surg. 2015 Oct;22:143-8. doi: 10.1016/j.ijsu.2015.08.033. Epub 2015 Aug 24. PMID 26316154